CLINICAL TRIAL: NCT06616467
Title: Cognitive-Behavioral Intervention Targeting Mothers to Increase Tummy Time Practice and Maintain Healthy Weight in Infants
Brief Title: Cognitive-Behavioral Intervention to Increase Tummy Time Practice and Maintain Healthy Weight in Infants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Collaborators: Universidad de la Sabana (Other)
Responsible Party: Principal Investigator, Gabriela Iveth Martínez Figueroa, Master in Nursing, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FAEN-D-2016
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Obesity/therapy; Prevention and Control
Keywords: Infants; Prone position; Health Behavior; Mothers
MeSH Terms: conditions — Obesity; Health Behavior

STUDY DESIGN:
Intervention Model Description: The present research will be a phase II intervention study (Gitlin & Czaja, 2016), of the Pilot Randomized Clinical Trial (RCT) type, because it is intended to manipulate the independent variable that will be the intervention that integrates the components of: knowledge, beliefs, infant temperament, self-efficacy and sedentary practices, to measure the effect on the variables dependent on Tummy Time practice practice and healthy weight control. The Experimental Group (EG) and Control Group (CG) will be randomized, the intervention will be with a single-blind approach and repeated measurements (Grove & Burns, 2015).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tummy Time Group (Experimental): This group will receive the 12-week intervention, which will have follow-up measurements during the implementation of the intervention.
  Interventions: Behavioral: Tummy Time for the prevention of childhood obesity
- Hospital Group (No Intervention): This group receives the usual hospital care where the mother is provided with general information on breastfeeding, vaccination and infant screening.

INTERVENTIONS:
Behavioral: Tummy Time for the prevention of childhood obesity — A cognitive-behavioral intervention aimed at mothers of infants is presented that aims to increase the practice of TT and maintain a healthy weight in the infant, called "Tummy Time for the prevention of childhood obesity", within the intervention modifiable variables are involved that directly impact the expected results such as: the knowledge and beliefs of the mothers, infant temperament, parental self-efficacy and self-efficacy for the practice of TT.
  The intervention lasts 12 weeks from the first contact with the participants and consists of eight sessions broken down as follows: the first session is presented in a face-to-face format with expository, audiovisual and demonstrative means; sessions two, four, five and seven are provided through a text message with use WhatsApp® and the use of visual media. Sessions three, six and eight are delivered via telephone call with the aim of offering feedback on the doubts generated up to that point.
  Arms: Tummy Time Group

SUMMARY:
Childhood obesity is a serious health problem worldwide evidenced by its high prevalence, specifically for the age group called the first 1000 days of life. This condition has serious consequences on the health of infants who suffer from it, being a precursor for the development of diseases such as diabetes and hypertension. For this reason, international organizations have proposed physical activity as a priority component for the prevention of childhood obesity. The objective of this study is to evaluate the preliminary effect of an intervention based on social cognitive theory aimed at Mexican mothers with children under six months of age to increase the practice of Tummy Time and maintain the healthy weight of the infant compared to usual care. The methodology will be a pilot randomized clinical trial with randomization to the Experimental Group and Control Group, the intervention will be with a single-blind approach and repeated measurements. A non-probabilistic sampling will be used for convenience and the sample will be 144 participants who will be dyads of mothers and children who are in the immediate postpartum hospitalized in a second-level hospital in Mexico.

ELIGIBILITY:
Inclusion Criteria:

* Mother-child dyads that are in the postpartum
* mothers who declare that they know how to read and write in spanish
* have an electronic device (cell phone, tablet or computer),
* have an internet connection.
* Have the social network WhatsApp®
* Agree to participate voluntarily evidenced by informed consent will be considered

Exclusion Criteria:

* Women who report having received information about TT one month before the intervention.
* Women who are actively participating in programs related to early stimulation
* Who declare that they have a premature infant born before 37 SDG,
* who has a low birth weight <2,500g,
* who has a medical condition or complication at birth that impacts their physical mobility and
* who has chronic health problems or congenital anomalies.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Increased practice of tummy time in infants | It will be measured at baseline, 3 and 6 months.
  The diary is made up of 15 items aimed at measuring whether the activity is applied, frequency with which it is performed, duration in each frequency and total duration of the activity within 24 hours, it is made up of open responses and must be answered according to the last week prior to the application of the instrument. The interpretation is made for each item and is compared with the recommendations given in the guidelines of international organizations (PAHO, 2019), the results are presented in a comparison to determine whether or not the recommendations given are complied with.
Maintenance of healthy weight in the infant | It will be measured at baseline, at 3 and 6 months of age of the infant.
  , the infant growth patterns in children under two years of age will be used, where the anthropometric measurements of infants during birth will be used and in the follow-up measurements self-reported by the mother, the data will be analyzed through the free access computer program Anthro ® of the WHO (2024) that allows calculating through the indicators of weight/length and BMI/age the nutritional status of the infant and be classified using the z-scores: malnutrition (≤ -2 SD); normal (≥ -1 and ≤ 1 SD); SP (> 1 and ≤ 2 DE) and OB (≥ 2 DE).

SECONDARY OUTCOMES:
increasing mothers' knowledge of developmental milestones | It will be measured at baseline, at 3 and 6 months
  The questionnaire "parents' knowledge of developmental milestones in children", developed and validated by Rickhy et al. (2010) in English, will be used, which aims to assess parents' knowledge about the time in which their children should achieve different skills. It consists of 17 questions distributed in five dimensions: 1) physical development (1, 2, 3 and 4); 2) cognitive development (5, 6 and 7); 3) social development (8, 9, 10, 11 and 12) and 4) and emotional development (13, 14, 15, 16 and 17), with a dichotomous response scale of 1= true, 2= false. For interpretation, the answers are graded at 1 = correct and 0 = incorrect, the score ranges from 0 to 17 points, it being understood that the higher the score, the higher the level of knowledge the parents have.
Increased knowledge of tummy time | Measured at baseline, 3 months and 6 months
  The questionnaire "knowledge, beliefs and implementation on the prone position" This indicator was developed and validated by Ricard and Metz (2014) in English, It consists of three dimensions, the first dimension measures knowledge about TT, it is made up of nine questions that are answered on a dichotomous scale of 1= true; 2= false, presented a Cronbach's alpha reliability of .67. For their interpretation, the questions are evaluated and transformed into 1= correct; 0= incorrect, the score ranges from 0 to 9 points, where it is interpreted that the higher the score, the higher the level of knowledge about TT the parents have.
Positive and negative beliefs about tummy time | Measured at baseline, 3 months and 6 months
  The questionnaire knowledge, beliefs and implementation on the prone position. This indicator was developed and validated by Ricard and Metz (2014) in English, It consists of three dimensions, The second dimension assesses parents' beliefs about TT is made up of 18 items with a five-point Likert-type response scale (1=strongly disagree, 2=disagree, 3=neither disagree nor agree, 4=agree and 5=strongly agree), is subdivided into positive beliefs (10, 11, 12, 13, 14, 15, 16, 17, and 18) and negative beliefs (1, 2, 3, 4, 5, 6, 7, 8, and 9), the questionnaire as a whole presented a Cronbach's alpha reliability of .45 in the original language; The total score ranges from 18 to 90 points, it is interpreted that the higher the score, the higher the level of positive and/or negative beliefs
increased implementation of tummy time | Measured at baseline, 3 months and 6 months
  The questionnaire knowledge, beliefs and implementation on the prone position. This indicator was developed and validated by Ricard and Metz (2014) in English, It consists of three dimensions, dimension three evaluates the factors, frequency and duration of TT in the infant, it is made up of 11 items with a multiple response scale for each item, the interpretation is descriptive per item.
Maternal Perception of Child's Weight | will be measured at baseline, 3 months and 6 months
  It is made up of an item of: "I think my child is" with a multiple choice of: underweight, a little underweight, more or less with the correct weight, with a little SP and with SP, it is also evaluated with a panel of five images according to the sex of the child, in which the mother must select two things: 1) the image that best represents the weight of her child and 2) the image that represents a healthy child. The selection of the answers will determine the mother's perception of her child's weight and a healthy weight.
Child Behavior | will be measured at baseline, 3 months and 6 months
  the questionnaire aims to measure infant temperament as a sign of the frequency in which the infant presents the behavior during a week prior to application. It is composed of 37 items with a 7-point Likert-type response scale ranging from 1= never to 7= always, and is divided into three dimensions. For the interpretation, item 11 evaluates inversely, a sum of the total of the items is made, where the total score ranges from 37 to 259 points, it is considered that, the higher the score, the greater the characteristic of infant temperament as a function of the three dimensions.
  Likewise, a subscale of "calming techniques" is presented, which aims to determine which techniques the mother has used to calm her child in the last two weeks, it is composed of 11 items with a 7-point Likert-type response scale ranging from 1= none to 7= always. The interpretation is carried out in a descriptive way of each item.
increased mother's self-confidence in child rearing | will be measured at baseline, 3 months and 6 months
  the "Karitane Parental Confidence Scale". It is composed of three dimensions of: 1) perceptions of parenting capacity; 2) available parenting support and 3) perceptions of child development. It is made up of a total of 15 items with a four-point Likert-type response scale of: 0 = No, almost never, 1 = No, not very often, 2 = Yes, sometimes, 3 = Yes, most of the time, with a range of scores from 0 to 45 maximum. The interpretation is made with the total sum of the items, where the higher the score, the higher the level of self-efficacy perceived by the parents for upbringing, in addition cohorts are presented according to the score where they have: severe clinical range (31 or less); moderate clinical range (31-35); mild clinical range (36-39) and no clinical range (40 or more).
Perceived Parental Self-Efficacy for Physical Activity Behaviors | will be measured at baseline, 3 months and 6 months
  the questionnaire "perceived parental self-efficacy on dietary and physical activity behavior", developed and validated by Bohman et al. (2013) in its English version. It is made up of 14 items that are subdivided into two dimensions: 1) self-efficacy for dietary behaviors (1, 2, 3, 4, 5, 6 and 7) and 2) self-efficacy for physical activity behaviors (8, 9, 10, 11, 12, 13 and 14), an 11-point Likert-type response scale ranging from 0= nothing to 10= to a very high degree, with a score ranging from 0 to 140, it is interpreted that, the higher the score, the greater the parents' perception of self-efficacy. It has presented reliability through Cronbach's alpha coefficient of .88.

CONTACTS AND LOCATIONS:
Overall Officials: Velia M Cárdenas Villarreal, PhD, Study Director — Universidad Autonoma de Nuevo León; Jorge A Mayo Abarca, Master, Study Chair — Universidad Autonoma de Nuevo León; Gloria Carvajal Carrascal, PhD, Study Chair — Universidad de la Sabana
Locations (1):
- Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No
Not due to the protection of participant confidentiality given by informed consent. Statistical data only.

REFERENCES:
- [Background] Taylor BJ, Heath AL, Galland BC, Gray AR, Lawrence JA, Sayers RM, Dale K, Coppell KJ, Taylor RW. Prevention of Overweight in Infancy (POI.nz) study: a randomised controlled trial of sleep, food and activity interventions for preventing overweight from birth. BMC Public Health. 2011 Dec 19;11:942. doi: 10.1186/1471-2458-11-942. PMID 22182309
- [Background] Taj F, Klein MCA, van Halteren A. Digital Health Behavior Change Technology: Bibliometric and Scoping Review of Two Decades of Research. JMIR Mhealth Uhealth. 2019 Dec 13;7(12):e13311. doi: 10.2196/13311. PMID 31833836
- [Background] Rosenstock S, Ingalls A, Foy Cuddy R, Neault N, Littlepage S, Cohoe L, Nelson L, Shephard-Yazzie K, Yazzie S, Alikhani A, Reid R, Kenney A, Barlow A. Effect of a Home-Visiting Intervention to Reduce Early Childhood Obesity Among Native American Children: A Randomized Clinical Trial. JAMA Pediatr. 2021 Feb 1;175(2):133-142. doi: 10.1001/jamapediatrics.2020.3557. PMID 33165594
- [Background] Rikhy S, Tough S, Trute B, Benzies K, Kehler H, Johnston DW. Gauging knowledge of developmental milestones among Albertan adults: a cross-sectional survey. BMC Public Health. 2010 Apr 8;10(1):183. doi: 10.1186/1471-2458-10-183. PMID 20377910
- [Background] Putnam SP, Helbig AL, Gartstein MA, Rothbart MK, Leerkes E. Development and assessment of short and very short forms of the infant behavior questionnaire-revised. J Pers Assess. 2014;96(4):445-58. doi: 10.1080/00223891.2013.841171. Epub 2013 Nov 9. PMID 24206185
- [Background] Poitras VJ, Gray CE, Janssen X, Aubert S, Carson V, Faulkner G, Goldfield GS, Reilly JJ, Sampson M, Tremblay MS. Systematic review of the relationships between sedentary behaviour and health indicators in the early years (0-4 years). BMC Public Health. 2017 Nov 20;17(Suppl 5):868. doi: 10.1186/s12889-017-4849-8. PMID 29219092
- [Background] Perez-Herrera A, Cruz-Lopez M. [Childhood obesity: current situation in Mexico]. Nutr Hosp. 2019 Apr 10;36(2):463-469. doi: 10.20960/nh.2116. Spanish. PMID 30866635
- [Background] Paul IM, Savage JS, Anzman-Frasca S, Marini ME, Beiler JS, Hess LB, Loken E, Birch LL. Effect of a Responsive Parenting Educational Intervention on Childhood Weight Outcomes at 3 Years of Age: The INSIGHT Randomized Clinical Trial. JAMA. 2018 Aug 7;320(5):461-468. doi: 10.1001/jama.2018.9432. PMID 30088009
- [Background] Palmer CF, Rindler D, Leverone B. Moving into tummy time, together: Touch and transitions aid parent confidence and infant development. Infant Ment Health J. 2019 Mar;40(2):277-288. doi: 10.1002/imhj.21771. Epub 2019 Jan 25. PMID 30681173
- [Background] Nitsos A, Estrada RD, Messias DKH. Tummy Time for Latinos With Limited English Proficiency: Evaluating the Feasibility of a Cultural and Linguistically Adapted Parent Education Intervention. J Pediatr Nurs. 2017 Sep-Oct;36:31-36. doi: 10.1016/j.pedn.2017.04.004. Epub 2017 May 17. PMID 28888509
- [Background] Michie S, Ashford S, Sniehotta FF, Dombrowski SU, Bishop A, French DP. A refined taxonomy of behaviour change techniques to help people change their physical activity and healthy eating behaviours: the CALO-RE taxonomy. Psychol Health. 2011 Nov;26(11):1479-98. doi: 10.1080/08870446.2010.540664. Epub 2011 Jun 28. PMID 21678185
- [Background] Michie S, Yardley L, West R, Patrick K, Greaves F. Developing and Evaluating Digital Interventions to Promote Behavior Change in Health and Health Care: Recommendations Resulting From an International Workshop. J Med Internet Res. 2017 Jun 29;19(6):e232. doi: 10.2196/jmir.7126. PMID 28663162
- [Background] McMillan AG, May LE, Gaines GG, Isler C, Kuehn D. Effects of Aerobic Exercise during Pregnancy on 1-Month Infant Neuromotor Skills. Med Sci Sports Exerc. 2019 Aug;51(8):1671-1676. doi: 10.1249/MSS.0000000000001958. PMID 30817721
- [Background] McEachan RRC, Santorelli G, Bryant M, Sahota P, Farrar D, Small N, Akhtar S, Sargent J, Barber SE, Taylor N, Richardson G, Farrin AJ, Bhopal RS, Bingham DD, Ahern SM, Wright J; BiB childhood obesity scientific group. The HAPPY (Healthy and Active Parenting Programmme for early Years) feasibility randomised control trial: acceptability and feasibility of an intervention to reduce infant obesity. BMC Public Health. 2016 Mar 1;16:211. doi: 10.1186/s12889-016-2861-z. PMID 26931491
- [Background] Mailhot T, Goulet MH, Maheu-Cadotte MA, Fontaine G, Lequin P, Lavoie P. Methodological reporting in feasibility studies: a descriptive review of the nursing intervention research literature. J Res Nurs. 2020 Aug;25(5):460-472. doi: 10.1177/1744987119883404. Epub 2019 Nov 26. PMID 34394661
- [Background] Lopez-Sobaler AM, Aparicio A, Salas-Gonzalez MD, Loria Kohen V, Bermejo Lopez LM. [Childhood obesity in Spain and associated factors]. Nutr Hosp. 2021 Sep 30;38(Spec No2):27-30. doi: 10.20960/nh.03793. Spanish. PMID 34323095
- [Background] Koren A, Kahn-D'angelo L, Reece SM, Gore R. Examining Childhood Obesity From Infancy: The Relationship Between Tummy Time, Infant BMI-z, Weight Gain, and Motor Development-An Exploratory Study. J Pediatr Health Care. 2019 Jan;33(1):80-91. doi: 10.1016/j.pedhc.2018.06.006. Epub 2018 Aug 18. PMID 30131199
- [Background] Korczak DJ, Madigan S, Colasanto M, Szatmari P, Chen Y, Maguire J, Parkin P, Birken CS. The longitudinal association between temperament and physical activity in young children. Prev Med. 2018 Jun;111:342-347. doi: 10.1016/j.ypmed.2017.11.021. Epub 2017 Nov 29. PMID 29197529
- [Background] Kieslinger K, Wartha O, Pollatos O, Steinacker JM, Kobel S. Parental Self-Efficacy-A Predictor of Children's Health Behaviors? Its Impact on Children's Physical Activity and Screen Media Use and Potential Interaction Effect Within a Health Promotion Program. Front Psychol. 2021 Aug 12;12:712796. doi: 10.3389/fpsyg.2021.712796. eCollection 2021. PMID 34456826
- [Background] Karimy M, Armoon B, Fayazi N, Koohestani HR. A Study on the Knowledge, Attitude, and Practices of Iranian Mothers towards Childhood Obesity. Obes Facts. 2019;12(6):669-677. doi: 10.1159/000492795. Epub 2019 Dec 16. PMID 31842015
- [Background] Jones RE, Jewell J, Saksena R, Ramos Salas X, Breda J. Overweight and Obesity in Children under 5 Years: Surveillance Opportunities and Challenges for the WHO European Region. Front Public Health. 2017 Apr 13;5:58. doi: 10.3389/fpubh.2017.00058. eCollection 2017. PMID 28451584
- [Background] Jia Z, Zhang J, Trindade D, Sobko T. Physical Activity Patterns and Correlates of 9-Month-Old Chinese Infants in the Macau Population. Matern Child Health J. 2018 Oct;22(10):1526-1533. doi: 10.1007/s10995-018-2614-y. PMID 30094531
- [Background] Hewitt L, Kerr E, Stanley RM, Okely AD. Tummy Time and Infant Health Outcomes: A Systematic Review. Pediatrics. 2020 Jun;145(6):e20192168. doi: 10.1542/peds.2019-2168. Epub 2020 May 5. PMID 32371428
- [Background] Hesketh KR, Janssen X. Movement behaviours and adherence to guidelines: perceptions of a sample of UK parents with children 0-18 months. Int J Behav Nutr Phys Act. 2022 May 21;19(1):58. doi: 10.1186/s12966-022-01300-5. PMID 35598015
- [Background] Hennessy M, Heary C, Laws R, van Rhoon L, Toomey E, Wolstenholme H, Byrne M. The effectiveness of health professional-delivered interventions during the first 1000 days to prevent overweight/obesity in children: A systematic review. Obes Rev. 2019 Dec;20(12):1691-1707. doi: 10.1111/obr.12924. Epub 2019 Sep 2. PMID 31478333
- [Background] Hemmingsson E. Early Childhood Obesity Risk Factors: Socioeconomic Adversity, Family Dysfunction, Offspring Distress, and Junk Food Self-Medication. Curr Obes Rep. 2018 Jun;7(2):204-209. doi: 10.1007/s13679-018-0310-2. PMID 29704182
- [Background] Haire-Joshu D, Tabak R. Preventing Obesity Across Generations: Evidence for Early Life Intervention. Annu Rev Public Health. 2016;37:253-71. doi: 10.1146/annurev-publhealth-032315-021859. PMID 26989828
- [Background] Gross RS, Mendelsohn AL, Yin HS, Tomopoulos S, Gross MB, Scheinmann R, Messito MJ. Randomized controlled trial of an early child obesity prevention intervention: Impacts on infant tummy time. Obesity (Silver Spring). 2017 May;25(5):920-927. doi: 10.1002/oby.21779. Epub 2017 Mar 22. PMID 28332324
- [Background] Galindo-Neto NM, Alexandre ACS, Barros LM, Sa GGM, Carvalho KM, Caetano JA. Creation and validation of an educational video for deaf people about cardiopulmonary resuscitation. Rev Lat Am Enfermagem. 2019 Mar 10;27:e3130. doi: 10.1590/1518-8345.2765.3130. PMID 30916231
- [Background] Flores-Pena Y, Aguado-Barrera ME, Cerda-Flores RM, Cortes-Gutierrez EI, Davila-Rodriguez MI. [Maternal perception of her child's weight and unrelated children less than 1 year old]. Aten Primaria. 2016 Nov;48(9):579-585. doi: 10.1016/j.aprim.2015.10.003. Epub 2015 Dec 22. Spanish. PMID 26718345
- [Background] Felzer-Kim IT, Erickson K, Adkins C, Hauck JL. Wakeful Prone "Tummy Time" During Infancy: How Can We Help Parents? Phys Occup Ther Pediatr. 2020;40(6):651-668. doi: 10.1080/01942638.2020.1742847. Epub 2020 Mar 19. PMID 32192403
- [Background] Estrada-Gutierrez G, Zambrano E, Polo-Oteyza E, Cardona-Perez A, Vadillo-Ortega F. Intervention during the first 1000 days in Mexico. Nutr Rev. 2020 Dec 1;78(Suppl 2):80-90. doi: 10.1093/nutrit/nuaa082. PMID 33196088
- [Background] Enright G, Allman-Farinelli M, Redfern J. Effectiveness of Family-Based Behavior Change Interventions on Obesity-Related Behavior Change in Children: A Realist Synthesis. Int J Environ Res Public Health. 2020 Jun 8;17(11):4099. doi: 10.3390/ijerph17114099. PMID 32521815
- [Background] Eichner-Seitz N, Pate RR, Paul IM. Physical activity in infancy and early childhood: a narrative review of interventions for prevention of obesity and associated health outcomes. Front Endocrinol (Lausanne). 2023 May 24;14:1155925. doi: 10.3389/fendo.2023.1155925. eCollection 2023. PMID 37293499
- [Background] Downing KL, Del Pozo Cruz B, Sanders T, Zheng M, Hnatiuk JA, Salmon J, Hesketh KD. Outdoor time, screen time and sleep reported across early childhood: concurrent trajectories and maternal predictors. Int J Behav Nutr Phys Act. 2022 Dec 29;19(1):160. doi: 10.1186/s12966-022-01386-x. PMID 36581865
- [Background] de Vries AG, Huiting HG, van den Heuvel ER, L'Abee C, Corpeleijn E, Stolk RP. An activity stimulation programme during a child's first year reduces some indicators of adiposity at the age of two-and-a-half. Acta Paediatr. 2015 Apr;104(4):414-21. doi: 10.1111/apa.12880. Epub 2015 Jan 7. PMID 25425024
- [Background] Dattilo AM, Saavedra JM. Nutrition Education: Application of Theory and Strategies during the First 1,000 Days for Healthy Growth. Nestle Nutr Inst Workshop Ser. 2019;92:1-18. doi: 10.1159/000499544. Epub 2019 Nov 28. PMID 31779004
- [Background] Wang Y, Min J, Khuri J, Li M. A Systematic Examination of the Association between Parental and Child Obesity across Countries. Adv Nutr. 2017 May 15;8(3):436-448. doi: 10.3945/an.116.013235. Print 2017 May. PMID 28507009
- [Background] Crncec R, Barnett B, Matthey S. Development of an instrument to assess perceived self-efficacy in the parents of infants. Res Nurs Health. 2008 Oct;31(5):442-53. doi: 10.1002/nur.20271. PMID 18297638
- [Background] Carson V, Zhang Z, Predy M, Pritchard L, Hesketh KD. Longitudinal associations between infant movement behaviours and development. Int J Behav Nutr Phys Act. 2022 Jan 28;19(1):10. doi: 10.1186/s12966-022-01248-6. PMID 35090492
- [Background] Carson V, Lee EY, Hewitt L, Jennings C, Hunter S, Kuzik N, Stearns JA, Unrau SP, Poitras VJ, Gray C, Adamo KB, Janssen I, Okely AD, Spence JC, Timmons BW, Sampson M, Tremblay MS. Systematic review of the relationships between physical activity and health indicators in the early years (0-4 years). BMC Public Health. 2017 Nov 20;17(Suppl 5):854. doi: 10.1186/s12889-017-4860-0. PMID 29219090
- [Background] Cardenas-Villarreal VM, Hernandez-Barrera L, Castro-Sifuentes D, Guevara-Valtier MC, Trejo-Valdivia B. Trends in overweight and obesity in children under 24 months of age in Mexico (2012-2020): analysis of four national health surveys. Cad Saude Publica. 2023 Dec 22;39(12):e00046123. doi: 10.1590/0102-311XEN046123. eCollection 2023. PMID 38126557
- [Background] Mendres-Smith AE, Borrero JC, Castillo MI, Davis BJ, Becraft JL, Hussey-Gardner B. Tummy time without the tears: The impact of parent positioning and play. J Appl Behav Anal. 2020 Sep;53(4):2090-2107. doi: 10.1002/jaba.715. Epub 2020 May 20. PMID 32436294
- [Background] Bohman B, Nyberg G, Sundblom E, Elinder LS. Validity and Reliability of a Parental Self-Efficacy Instrument in the Healthy School Start Prevention Trial of Childhood Obesity. Health Educ Behav. 2014 Aug;41(4):392-6. doi: 10.1177/1090198113515243. Epub 2013 Dec 25. PMID 24369178
- [Background] Black MM, Hager ER, Wang Y, Hurley KM, Latta LW, Candelaria M, Caulfield LE. Toddler obesity prevention: A two-generation randomized attention-controlled trial. Matern Child Nutr. 2021 Jan;17(1):e13075. doi: 10.1111/mcn.13075. Epub 2020 Sep 4. PMID 32885909
- [Background] Ardic C, Usta O, Omar E, Yildiz C, Memis E. Effects of infant feeding practices and maternal characteristics on early childhood obesity. Arch Argent Pediatr. 2019 Feb 1;117(1):26-33. doi: 10.5546/aap.2019.eng.26. English, Spanish. PMID 30652443
- [Background] Alves JGB, Alves GV. Effects of physical activity on children's growth. J Pediatr (Rio J). 2019 Mar-Apr;95 Suppl 1:72-78. doi: 10.1016/j.jped.2018.11.003. Epub 2018 Dec 26. PMID 30593790
- [Background] Alhwoaimel NA, Almarzoug H, Aldukhaini R, Altamimi R, Aldosre M, Al-Faris S, Azab AR. Parental knowledge of children's motor development: A cross-sectional study in Saudi Arabia. Res Dev Disabil. 2023 Aug;139:104552. doi: 10.1016/j.ridd.2023.104552. Epub 2023 Jun 7. PMID 37295126
- See also: Mexican Association of Market Intelligence and Opinion Agencies — https://www.amai.org/NSE/index.php
- See also: UNICEF Program Guide: Prevention of Overweight and Obesity in Children and Adolescents. — https://www.unicef.org/media/96096/file/Overweight-Guidance-2020-ES.pdf
- See also: Establishment of priority areas of action for the prevention of Childhood Obesity. — https://apps.who.int/iris/bitstream/handle/10665/250750/9789243503271-spa.pdf;sequence=1
- See also: Obesity and overweight. — https://www.who.int/es/news-room/fact-sheets/detail/obesity-and-overweight
- See also: WHO Child Growth Patterns: Training Course on Child Growth Assessment — https://www.paho.org/hq/dmdocuments/2009/Module_C_final.pdf
- See also: Regulation of the General Health Law on Health Research. DOF 02-04-2014 — https://www.diputados.gob.mx/LeyesBiblio/regley/Reg_LGS_MIS.pdf